CLINICAL TRIAL: NCT07330687
Title: A Brain Imaging Study of Abnormal Neural Network Reorganization Following Speech Training in Patients With Compensatory Articulation Secondary to Cleft Palate
Brief Title: Neural Changes After Speech Therapy in Patients With Cleft Palate: A Brain Imaging Study
Acronym: fMRI-Speech-CP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shufan Zhao (Other)
Collaborators: Guangzhou Women and Children's Medical Center (Other); Wenzhou Medical University (Other); National Natural Science Foundation of China (Other Government)
Responsible Party: Sponsor-Investigator, Shufan Zhao, PhD, Attending Physician, Wenzhou Medical University
Organization: Wenzhou Medical University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017021923
Record Dates: First submitted 2025-12-28; First posted 2026-01-09 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Cleft Lip and/or Palate; Speech Disorder; Speech Therapy; Brain; Magnetic Resonance Imaging
MeSH Terms: conditions — Speech Disorders; Communication Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Non-Oral Articulation(NOA) group (Experimental): Participants receive the investigational behavioral intervention: Structured Speech Decompensation Therapy. This one-on-one therapy uses the glottal stop /kʔ/ as a key sound to guide correct articulation placement and correct compensatory habits, integrating multisensory cues. The intervention is administered by a certified speech therapist at a dosage of 1-hour sessions, with a frequency of 3 sessions per week, for a duration of 5 to 12 weeks. Parent participation in sessions and daily prescribed home practice are required components.
  Interventions: Behavioral: Structured Speech Training for Decompensation
- Oral Articulation (OA) Group (No Intervention): Participants do not receive the investigational speech training intervention. This arm serves as the clinical control group.
- healthy control(HC) (No Intervention): Participants do not receive any study-related intervention. This arm serves as the healthy normative control group.

INTERVENTIONS:
Behavioral: Structured Speech Training for Decompensation — This structured, one-on-one speech decompensation therapy targets Non-oral Articulation Disorder (NOA) in postoperative cleft palate patients, using the glottal stop /kʔ/ as a key sound to guide correct articulation placement and correct compensatory habits. It follows a structured paradigm from error recognition to generalization, integrating multisensory cues. Delivered by a therapist 3 times/week for 1 hour over 5-12 weeks with parent participation, it includes daily home practice. Completion requires accurate sound production, with daily parent-supervised maintenance practice for one year thereafter.
  Arms: Non-Oral Articulation(NOA) group

SUMMARY:
Cleft palate is one of the most common maxillofacial congenital malformations, which results in severe speech disorders. Compensatory articulation disorder, also known as non-oral articulation disorder (NOA), is considered as the major pathological change among these patients. However, the outcome of speech therapy, an important treatment method, for NOA is often unsatisfactory. This is attributed to the erroneous articulation patterns and entrenched habits in patients with NOA, which require considerable training intensity and time. According to preliminary results from the investigators' own study, as well as studies by others, structural and functional changes have been clearly identified in some brain regions of patients with NOA, suggesting that abnormal neural networks are involved in the progression of NOA. Thus, the investigators proposed the hypothesis that speech therapy effectively corrects articulation disorders through reconfiguration of pathological neural function and reorganization of the abnormal neural network involved in NOA. In this study, multimodal brain imaging techniques will be applied to investigate differences in brain functional connectivity and structural connectivity networks among groups with oral articulation (OA), varying degrees of NOA in postoperative cleft palate patients, and healthy controls. The relationship between improvement in speech intelligibility and alterations in brain networks before and after intervention will be compared. This study aims to reveal the neural network substrates associated with NOA and speech therapy. Overall, through this comprehensive study, the investigators aim not only to provide new insight into the underlying neural mechanism of NOA but also to accumulate evidence for improving the efficacy of speech therapy and discovering new therapeutic strategies in clinical practice.

DETAILED DESCRIPTION:
Cleft palate often leads to compensatory articulation disorder (Non-oral Articulation, NOA), which is resistant to conventional speech therapy. This study is grounded in the hypothesis that the efficacy of speech training is mediated by the reorganization of pathological neural networks and structures associated with NOA.

This non-randomized, longitudinal study employs a parallel-group design involving three cohorts: patients with NOA receiving speech training, postoperative cleft palate patients with normal oral articulation (OA) as a clinical control, and healthy controls. The primary objective is to identify the distinctive neural signatures (in both functional connectivity and brain structure) linked to NOA and its remediation through training.

All participants undergo multimodal magnetic resonance imaging (including high-resolution T1-weighted and resting-state functional scans) and standardized speech assessments at baseline. Only the NOA group then receives a structured speech training intervention, followed by post-intervention reevaluation. By comparing changes within and between groups, this study aims to disentangle neural alterations specific to NOA from those related to cleft palate in general.

The integrative analysis of brain-wide changes with a focus on speech-related regions is expected to provide a systems-level understanding of the neural mechanisms underlying NOA and treatment-induced recovery. The findings may contribute to the development of more effective, neuroscience-informed therapeutic strategies.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 4 and 16 years.
* For patient groups: Diagnosed with non-syndromic cleft palate and having undergone cleft palate repair surgery at least 1 year prior.
* For the NOA group: Diagnosed with compensatory articulation disorder (Non-oral Articulation, NOA) through standardized speech assessment.
* For the OA group: Confirmed to have no compensatory articulation disorder (Oral Articulation, OA) through standardized speech assessment.
* For the healthy control group: No history of any craniofacial malformations, speech disorders, or neurological diseases.
* Participants and their legal guardians are able to understand and willing to provide written informed consent.
* Able to cooperate with and complete magnetic resonance imaging (MRI) examinations (e.g., no claustrophobia, no contraindicated metal implants).

Exclusion Criteria:

* Presence of other known syndromes or cognitive impairments (e.g., autism spectrum disorder, intellectual disability).
* History of other neurological diseases that may affect speech function (e.g., cerebral palsy, hearing loss).
* Presence of severe other orofacial anomalies, or an unrepaired palatal fistula.
* Contraindications for MRI examination (e.g., non-removable metal implants, severe claustrophobia).
* Having received systematic speech therapy within the past 6 months.
* Any other condition deemed by the investigator to be unsuitable for participation in the study.

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 164 (Actual)
Dates: Start 2019-01-06 (Actual); Primary Completion 2021-05-27 (Actual); Study Completion 2021-08-21 (Actual)

PRIMARY OUTCOMES:
Change in Functional Connectivity of the Speech Related Network | From baseline assessment to post-training assessment (approximately at Week 12)
  Change in resting-state functional connectivity, focusing on connections between pre-defined speech-related regions (Broca's and Wernicke's areas) and additionally assessed through whole-brain network analysis, using resting-state fMRI data.
Change in Percent Correct Consonants (PCC) | From baseline assessment to post-training assessment (approximately at Week 12)
  Change in the percentage of consonants produced correctly, assessed within both single-word and conversational speech contexts. The measure is derived from standardized speech samples, which are evaluated by blinded, certified speech-language pathologists.

SECONDARY OUTCOMES:
Change in Grey Matter Volume (GMV) of Articulation-Related Regions | From baseline to post-training assessment (at Week 12)
  Alterations in grey matter volume across the whole brain, with a focus on regions implicated in articulation. Measured by voxel-based morphometry (VBM) analysis of high-resolution T1-weighted magnetic resonance imaging (MRI) scans.
Change in Regional Homogeneity (ReHo) in Speech-Related Cortex | From baseline to post-training assessment (at Week 12)
  Changes in local brain activity synchronization across the whole brain, with particular emphasis on the speech-related cortex.
Change in Amplitude of Low-Frequency Fluctuations (fALFF) | From baseline to post-training assessment (at Week 12)
  Changes in the fractional amplitude of low-frequency fluctuations in the blood-oxygen-level-dependent (BOLD) signal across the whole brain, assessed within regions of the speech and auditory processing networks. Derived from resting-state fMRI data.
Change in Proportion of Compensatory Articulation Errors | From baseline to post-training assessment (at Week 12)
  Change in the proportion of compensatory (non-oral) articulation errors relative to the total number of consonants attempted, analyzed within both single-word and conversational speech samples. This metric is calculated through phonetic transcription of the speech samples to quantify the frequency of error patterns characteristic of non-oral articulation.
Change in White Matter Volume (WMV) of Articulation-Related Regions | From baseline to post-training assessment (at Week 12)
  Alterations in white matter volume across the whole brain, particularly within tracts associated with speech motor pathways. Analyzed using voxel-based analysis of T1-weighted MRI to quantify white matter volume changes.

CONTACTS AND LOCATIONS:
Locations (1):
- School & Hospital of Stomatology Wenzhou Medical University, Wenzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No
A final decision regarding the sharing of individual participant data (IPD) has not been made at the time of this registration. This study involves sensitive neuroimaging and speech data. Data sharing considerations, including the feasibility of complete de-identification, compliance with local regulations and ethical approvals, and the establishment of appropriate data access protocols, require further review by the study investigators and sponsoring institution. A formal data sharing plan may be developed in the future and will be made available upon reasonable request or via a controlled-access repository if deemed feasible and appropriate.

REFERENCES:
- [Result] Zhang W, Li C, Chen L, Xing X, Li X, Yang Z, Zhang H, Chen R. Increased activation of the hippocampus during a Chinese character subvocalization task in adults with cleft lip and palate palatoplasty and speech therapy. Neuroreport. 2017 Aug 16;28(12):739-744. doi: 10.1097/WNR.0000000000000832. PMID 28658048
- [Result] Wang Y, Deng C, Li H, Gao Y, Shi B, Huang X, Gong Q. Intranetwork and Internetwork Functional Connectivity Changes Related to Speech Disorders in Adults With Cleft Lip and Palate. Eur J Neurosci. 2025 Apr;61(7):e70077. doi: 10.1111/ejn.70077. PMID 40219708
- [Result] Zhang W, Guan Z, Cao L, Sun L, Zhang X, Chen R, Li C, Song W. Articulation-function-associated brain developmental changes in cleft lip and palate patients. Brain Res Bull. 2025 Sep;229:111458. doi: 10.1016/j.brainresbull.2025.111458. Epub 2025 Jul 11. PMID 40653058
- [Result] Zhang W, Zhao C, Sun L, Yang X, Yang L, Liang Y, Zhang X, Du X, Chen R, Li C. Articulation-Function-Associated Cortical Developmental Changes in Patients with Cleft Lip and Palate. Brain Sci. 2023 Mar 25;13(4):550. doi: 10.3390/brainsci13040550. PMID 37190514
- [Result] Wang S, Fang L, Miao G, Li Z, Rao B, Cheng H. Atypical cortical thickness and folding of language regions in Chinese nonsyndromic cleft lip and palate children after speech rehabilitation. Front Neurol. 2022 Sep 20;13:996459. doi: 10.3389/fneur.2022.996459. eCollection 2022. PMID 36203989
- [Result] Homoud NN, Ireland AJ, Sherriff M, AlSaffar Z, Davies AJV, Sandy JR. A Review and Meta-Analysis on Altered Brain Structure in Patients Born with Non-Syndromic Cleft Lip and/or Palate. Cleft Palate Craniofac J. 2025 Mar 24:10556656251327526. doi: 10.1177/10556656251327526. Online ahead of print. PMID 40129165